CLINICAL TRIAL: NCT00009555
Title: A Prospective, Multicenter, Randomized, Placebo-Controlled Trial of Physiologic Testosterone Supplementation for HIV-Positive Men With Mildly to Moderately Reduced Serum Testosterone Levels and Abdominal Obesity
Brief Title: Testosterone for HIV-Positive Men With Reduced Serum Testosterone Levels and Abdominal Fat
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: A5079; 10175 (Registry Identifier: DAIDS ES); ACTG A5079; AACTG A5079
Record Dates: First submitted 2001-02-01; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Testosterone; Anthropometry; Obesity; Abdomen
MeSH Terms: conditions — HIV Infections; Obesity | interventions — Testosterone

INTERVENTIONS:
Drug: Testosterone

SUMMARY:
The purpose of this study is to see if treatment with testosterone will reduce abdominal fat in HIV-positive men.

Many HIV patients on antiretroviral therapy show an increase in abdominal fat. Studies have shown that treatment with testosterone may decrease abdominal fat. This study will determine if testosterone will reduce abdominal fat in HIV patients.

DETAILED DESCRIPTION:
Reports suggest that many HIV-infected patients on antiretroviral therapy experience an increase in abdominal fat. The mechanisms of abdominal fat accumulation in HIV-infected patients are not known. Studies have shown: treatment with testosterone gel reduces total body fat in young, androgen-deficient men; testosterone replacement in middle-aged men with mid-segment obesity decreases visceral fat; and replacement doses of testosterone decrease fat mass and augment lean body mass in HIV-infected men with androgen deficiency. Therefore, there is a strong rationale for evaluating the effectiveness of testosterone replacement in HIV-infected men with visceral obesity and low testosterone levels.

Patients are stratified based on their viral load. Patients receive either testosterone gel or placebo applied to the skin once daily for 24 weeks. Patients remain on their current antiretroviral regimens, which are not supplied through the study. Patients who receive testosterone during the first 24 weeks are eligible to receive it for an additional 24 weeks. Patients on placebo are followed for an additional 24 weeks. Clinical and laboratory evaluations for visceral fat changes are performed throughout the study.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have been taking anti-HIV medications for at least 12 weeks before study entry and plan to continue taking them for an additional 24 weeks.
* Are male and between 18 and 70 years old.
* Have a measurement of greater than 100 cm around the abdomen.
* Can report an increase in abdominal size after taking antiretroviral drugs.
* Have a viral load less than 10,000 copies/ml within 6 weeks prior to screening.
* Have a serum total testosterone between 125 and 400 ng/dl. If serum total testosterone is greater than 400 ng/dl, bioavailable testosterone must be less than 115 ng/dl or free testosterone must be less than 50 pg/ml.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Take certain drugs, including testosterone derivatives, glucocorticoids, appetite stimulants, dronabinol, megestrol acetate, androstenediols, oxandrolone, or other anabolic agents such as dehydroepiandrosterone (DHEA) or growth hormone within 12 weeks prior to study entry.
* Take hydroxyurea within 30 days of study entry.
* Take drugs for diabetes.
* Have diabetes.
* Take granulocyte-macrophage colony-stimulating factor (GM-CSF). (Granulocyte colony-stimulating factor (G-CSF) is allowed.)
* Take cytokines, cytokine inhibitors, or ketoconazole.
* Take ritonavir with simvastatin or lovastatin.
* Have an active opportunistic infection. Patients on treatment for at least 12 weeks will be allowed.
* Have 5-7 loose stools per day or diarrhea for more than 1 week, within 6 weeks of study entry.
* Have a blood pressure greater than 160 over 100.
* Have certain heart problems.
* Have a breast mass that has not been diagnosed.
* Have active cancer.
* Have had prostate cancer or certain other prostate problems.
* Are allergic to any part of the testosterone gel.
* Have a history of blood clots.
* Have a history of sleep apnea.
* Are receiving experimental treatment.
* Are receiving experimental drugs in other studies and do not know if they are taking the drug or placebo.
* Abuse drugs or alcohol in a way that would interfere with the study.
* Are dieting or doing heavy exercising.
* Have a viral load of 10,000 copies/ml or more at screening

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86
Dates: Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shalender Bhasin, Study Chair; Cecilia Shikuma, Study Chair
Locations (27):
- United States (26):
  - USC CRS, Los Angeles, California
  - Charles R. Drew Univ. of Medicine and Science, Div. of Infectious Diseases, Los Angeles, California
  - Stanford CRS, Palo Alto, California
  - Ucsd, Avrc Crs, San Diego, California
  - Ucsf Aids Crs, San Francisco, California
  - Santa Clara Valley Med. Ctr., San Jose, California
  - San Mateo County AIDS Program, San Mateo, California
  - Marin County Dept. of Health & Human Services, HIV/AIDS Program & Specialty Clinic, San Rafael, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Queens Med. Ctr., Honolulu, Hawaii
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Northwestern University CRS, Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Indiana Univ. School of Medicine, Wishard Memorial, Indianapolis, Indiana
  - Methodist Hosp. of Indiana, Indianapolis, Indiana
  - IHV Baltimore Treatment CRS, Baltimore, Maryland
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - Washington U CRS, St Louis, Missouri
  - Univ. of Nebraska Med. Ctr., Durham Outpatient Ctr., Omaha, Nebraska
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - Univ. of Pennsylvania Health System, Presbyterian Med. Ctr., Philadelphia, Pennsylvania
  - Pitt CRS, Pittsburgh, Pennsylvania
- Puerto Rico-AIDS CRS, San Juan, Puerto Rico